

## **Statistical Analysis Plan**

## **Study Title:**

An investigation into neuropilates on motor function in chronic stroke: a pilot randomised feasibility study

**Document creation date:** August 4<sup>th</sup> 2020

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]



## **Statistical Analysis**

We will analyse the data using Excel and SPSS for Windows. Paired T tests will be used to compare before and after data in both groups.